CLINICAL TRIAL: NCT01679912
Title: Hereditary Angioedema : Interest From the Use of a Call Center During the Attacks.
Brief Title: A Call Center During HAE Attacks (SOS HAE)
Acronym: SOS AOH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110109; 2012-A00044-39 (Other: IDRCB)
Record Dates: First submitted 2012-08-21; First posted 2012-09-06 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; Emergency Medical Service; Health care coast; Telephone
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: phone to call center (Experimental): recommendations to phone to the call center for all the patients who have an acute attack
  Interventions: Other: phone to the call center
- 2: usual strategy (No Intervention): usual strategy. No intervention (patients does not change their practice)

INTERVENTIONS:
Other: phone to the call center — recommendations to phone to the call center for all the patients who have an acute attack
  Arms: 1: phone to call center

SUMMARY:
This clinical trial aims to compare morbidity and cost associated with acute attacks of hereditary angioedema in patients with an intervention based on a support after a phone call to the call center (SOS HAE) from a group of patients does not change their practice.

DETAILED DESCRIPTION:
Investigators propose a study to determine whether a call center for an acute attack of HAE associated with intervention recommendations based on systematic early treatment (self-administration at home or by a caregiver) would reduce the morbidity and the socioeconomic impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an hereditary angioedema followed in a reference center for bradykinin angioedema (CRéAk)
* Patient's age ≥ 18 years
* Consent to the participation in the study
* Affiliated to social security

Exclusion Criteria:

* pregnant woman
* recent history of myocardial infarction
* recent history of stroke
* allergy to icatibant or C1 inhibitor concentrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of hospital admissions for angioedema attack- no (%) | at 2 years

SECONDARY OUTCOMES:
Number of ICU admissions - no (%) | at 2 years
Number of ED admissions - no (%) | at 2 years
Number of hospital admissions for others causes - no (%) | at 2 years
Number of intubations - no (%) | at 2 years
Number of EMS interventions - no (%) | at 2 years
Number of working days lost | at 2 years
Mortality - no (%) | at 2 years
Mortality for angioedema attack- no (%) | at 2 years
Cost of angioedema attacks | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ADNET, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SAMU 93 - Hôpital Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Javaud N, Altar A, Fain O, Reuter PG, Desmaizieres M, Petrovic T, Ghazali A, Durand-Zaleski I, Bouillet L, Vicaut E, Launay D, Martin L, Floccard B, Gompel A, Sobel A, Boccon-Gibod I, Kanny G, Lapostolle F, Adnet F. Hereditary angioedema, emergency management of attacks by a call center. Eur J Intern Med. 2019 Sep;67:42-46. doi: 10.1016/j.ejim.2019.05.007. Epub 2019 May 18. PMID 31109849
- [Derived] Javaud N, Fain O, Durand-Zaleski I, Launay D, Bouillet L, Gompel A, Sobel A, Woimant M, Rabetrano H, Petrovic T, Lapostolle F, Boccon-Gibod I, Reuter PG, Bertrand P, Mezaour M, Coppere B, Floccard B, Kanny G, Baker E, Martin L, Vicaut E, Adnet F. Specialist Advice Support for Management of Severe Hereditary Angioedema Attacks: A Multicenter Cluster-Randomized Controlled Trial. Ann Emerg Med. 2018 Aug;72(2):194-203.e1. doi: 10.1016/j.annemergmed.2018.01.053. Epub 2018 Mar 2. PMID 29503044
- [Derived] Javaud N, Fain O, Durand-Zaleski I, Launay D, Bouillet L, Gompel A, Sobel A, Woimant M, Rabetrano H, Petrovic T, Lapostolle F, Boccon-Gibod I, Reuter PG, Bertrand P, Coppere B, Floccard B, Kanny G, Martin L, Vicaut E, Adnet F. Dedicated call center (SOS-HAE) for hereditary angioedema attacks: study protocol for a randomised controlled trial. Trials. 2016 Apr 30;17(1):225. doi: 10.1186/s13063-016-1350-0. PMID 27140403